CLINICAL TRIAL: NCT05458154
Title: Evaluation and Re-evaluation of Post-mastectomy Pain Syndrome by Breast Cancer EDGE Task Force Outcomes: Clinical Measures of Pain After Pain Management Protocol of Physiotherapy
Brief Title: Evaluation and Re-evaluation of Post-mastectomy Pain Syndrome by Breast Cancer EDGE Task Force Outcomes
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: General Committee of Teaching Hospitals and Institutes, Egypt (Other Government)
Responsible Party: Principal Investigator, Omnia Saeed Mahmoud Ahmed, Lecturer of Physical therapy, General Committee of Teaching Hospitals and Institutes, Egypt
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 202103030005
Record Dates: First submitted 2022-06-29; First posted 2022-07-14 (Actual); Last update posted 2022-07-14 (Actual); Status verified 2022-07

CONDITIONS: Post-mastectomy Pain Syndrome
Keywords: breast cancer; mastectomy; pain; syndrome; Assessment; EDGE task force; physiotherapy
MeSH Terms: conditions — Breast Neoplasms; Pain; Syndrome | interventions — Surveys and Questionnaires

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Experimental group (Experimental): Seven of the 22 pain measures demonstrated satisfactory psychometric properties and clinical utility and are thereby recommended for clinical and research use in adults with a diagnosis of cancer.
  Participants received Physical therapy program is critical to preserve flexibility, strength, range of motion, and normal neuromuscular recruitment. Patients' efforts to cut back their pain through avoidance behaviors can severely undermine function if mobility, activity of daily living, performance, or vocational capacity are affected. Physical therapy may involve trials of analgesic modalities like desensitization techniques, transcutaneous electrical nerve stimulation (TENS), and topical cold. Modality trials are rapid, relatively harmless, and inexpensive with the additional benefit that patients can self-administer effective treatments The pain management protocol of physiotherapy of PMPS depends mainly on education regarding the subsequent points that are paramount.
  Interventions: Other: questionnaires

INTERVENTIONS:
Other: questionnaires — Participants were recruited from the Baheya Centre for Early Detection and Treatment of Breast Cancer institution. Patients were eligible if they had a previously post-mastectomy pain syndrome (PMPS), and were presented with pain within the surgical area lasting more than 3 months. They were evaluated by questionnaires and methods of pain assessment then received their physiotherapy program specific for pain relief for six sessions, and so re-evaluation. All women gave informed written consent in Arabic and English forms.

SUMMARY:
The purpose of the Breast Cancer EDGE Task Force is to provide physiotherapists with a comprehensive list of outcome measures that can be administered to a selected patient population, to assess post-mastectomy pain syndrome.

DETAILED DESCRIPTION:
Female breast cancer incidence rates are slowly increasing by about 0.5% each year since the mid-2000s, attributed a minimum of partially to continued declines in fertility and increases in excess weight. the best number of deaths are from cancers of the lung, prostate, and colorectum in men and of the lung, breast, and colorectum in women. Incidence from 2014 through 2018 continued a slow increase for female breast cancer. For women, breast cancer, and lung cancer, account for 51% of all new diagnoses, with breast cancer alone accounting for nearly one-third.

According to the literature, the prevalence of chronic pain after breast cancer treatment varies from 25% to 60% in other countries.

Survival rates for breast cancer vary worldwide, but normally, rates have improved. In most countries, the five-year survival rate of early-stage breast cancers is 80-90 percent, falling to 24 percent for breast cancers diagnosed at a more advanced stage.

A systematic review evaluating risk factors for the event of persistent pain after surgery found that additionally to younger age, preoperative pain, intercostobrachial nerve damage during surgery, radiotherapy, also psychological morbidities are among the foremost frequently reported factors associated with chronic pain after breast cancer treatment.

Surgery could be a mainstay of primary breast cancer therapy. Alterations in surgical technique have reduced normal tissue injury, yet pain and functional compromise continue to occur following treatment.

Assa suggested that damage to the intercostobrachial nerve (ICBN) is also chargeable for the event of persistent pain arises from the lateral cutaneous branch of the second intercostal nerve and enters the axilla by perforating the second intercostal space and musculus serratus anterior within the midaxillary line. It then passes with considerable variability to the posteromedial border of the upper arm, leaving the ICBN in danger of harm during axillary surgery Post-mastectomy pain syndrome (PMPS) could be a chronic pain condition, typically neuropathic, which might occur following surgery on the breast.

Pain may be a common complication of breast cancer surgery. The event of chronic pain is one of the foremost frequently seen sequelae within the cancer survivor population.

Persistent pain after mastectomy was first reported during the 1970s, characterized as a dull, burning, and aching sensation within the anterior chest, arm, and axilla, exacerbated by movement of the shoulder girdle.

Although the pain related to breast cancer surgery includes different conditions (e.g., phantom-breast pain, pain around the mastectomy scar, or pain within the anterior chest wall). neuropathic pain due to intercostobrachial neuropathy-i.e. painful intercostobrachial neuropathy-is the foremost representative type of pain in breast cancer survivors The exact explanation for PMPS is unclear, but various etiological theories are postulated, including dissection of the intercostobrachial nerve, intraoperative damage to axillary nerve pathways, and pain caused by a neuroma, although evidence regarding the epidemiology of PMPS is growing, little is known about risk factors for the event of PMPS, or the long-term outcome of this chronic pain condition.

the International Association for the Study of Pain has defined chronic pain as that persisting beyond the traditional healing time of three months. Chronic pain was defined as PMPS supported by three criteria: character, location, and timing of pain. The identical criteria for PMPS were used at both time points to make sure comparability. Pain location was recorded as the same side of surgery, chest wall, axilla, or ipsilateral arm.

And "unpleasant sensory and emotional experience related to actual or potential tissue damage, or described in terms of such damage".

As the lesion recovers or the threat disappears, the pain sensation should normally decrease. However, when the pain remains persistent after the traditional tissue healing process, it can be considered chronic.

But, Neuropathic pain (NP), is defined by the International Association for the Study of Pain (IASP) as ''pain arising as a direct consequence of a lesion or disease affecting the somatosensory system will be a vital source of disability and distress in breast cancer patients already laid low with the psychological and medical stressors related to diagnosis and treatment and has been considered the foremost important contributor to chronic breast pain.

Neuropathic pain following breast surgery is often characterized by radiating pain, numbness, pins, and needles, burning, or stabbing. and is often related to paresthesia and hypersensitivity near the operative site.

The development of postoperative neuropathic pain (NPP) is related to many psychosocial and medical stressors, and for several, it represents a failure to return to normal life The current literature shows that chronic pain is related to nerve damage associated with the surgical technique, adjuvant therapy (such as chemotherapy, radiotherapy, and endocrine therapy), and younger age. However, these findings are equivocal because there's a body of literature that found no association between chemotherapy and chronic pain.

An important portion of breast cancer survivors needs to cope with complications and sequelae physical (lymphedema, neuropathy/pain, fatigue, menopausal symptoms, weight gain, etc.) and psychological nature (fear of recurrence, fear of death, change in body image, change in relationship, financial stress, etc.). These complications can arise during the treatment or can persist long after treatment cessation.

ELIGIBILITY:
Inclusion Criteria:

* Chronic pain >= 3 months
* Pain is localized to the chest wall or axilla.
* The onset of pain is clearly after surgery or radiation therapy.
* Pain is persistent, not fluctuating.
* The patient is a minimum of 6 weeks post-radiation therapy.

Exclusion Criteria:

* Time since surgery was less than 6 months.
* The pain wasn't presented as an outcome, previous ipsilateral breast cancer, pregnancy, disease within the nervous system, psychiatric disease.
* Time since diagnosis was less than 1 year.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 10 (Actual)
Dates: Start 2021-03-03 (Actual); Primary Completion 2022-03-03 (Actual); Study Completion 2022-04-04 (Actual)

PRIMARY OUTCOMES:
McGill Pain Questionnaire-Short Form | baseline
  15-word descriptors that describe two dimensions of pain: sensory and affective.
Numeric Rating Scale | baseline
  the most ordinarily used one is the 11-item version, the rating of pain from (0 - 10).
Visual Analog Scale | baseline
  is a 10 cm-long horizontal line with the words "no pain" at one end and "pain as bad as it can be" at the other.

SECONDARY OUTCOMES:
Brief Pain Inventory | baseline
  There's a complete of 32 items on the Brief Pain Inventory, it describes pain interferes with 7 domains of function within the last 24 hours:
  general activity, mood, walking ability, normal work, relations with people, sleep, and pleasure of life using a scale from 0 (no pain) to 10 (pain as bad as you can imagine).
Brief Pain Inventory-Short Form | baseline
  is a tool developed specifically to be used in individuals with cancer.
McGill Pain Questionnaire | baseline
  is a unique measure because it assesses pain using a multidimensional approach based on the gate control theoretical framework.
  contains three major classes of word descriptors: sensory, affective, and evaluative.
Pain Disability Index | baseline
  is a multidimensional tool designed to measure the degree to of chronic pain affects an individual's ability to perform a variety of activities.
  The PDI contains seven categories: family/home responsibility, recreation, social activity, occupation, sexual behavior, self-care, and life support activity.

CONTACTS AND LOCATIONS:
Locations (1):
- Baheya Centre for Early Detection and Treatment of Breast Cancer institution, Giza, Haram, Egypt

REFERENCES:
- [Background] Siegel RL, Miller KD, Fuchs HE, Jemal A. Cancer statistics, 2022. CA Cancer J Clin. 2022 Jan;72(1):7-33. doi: 10.3322/caac.21708. Epub 2022 Jan 12. PMID 35020204
- [Background] Kudel I, Edwards RR, Kozachik S, Block BM, Agarwal S, Heinberg LJ, Haythornthwaite J, Raja SN. Predictors and consequences of multiple persistent postmastectomy pains. J Pain Symptom Manage. 2007 Dec;34(6):619-27. doi: 10.1016/j.jpainsymman.2007.01.013. Epub 2007 Jul 16. PMID 17629668
- [Background] Poleshuck EL, Katz J, Andrus CH, Hogan LA, Jung BF, Kulick DI, Dworkin RH. Risk factors for chronic pain following breast cancer surgery: a prospective study. J Pain. 2006 Sep;7(9):626-34. doi: 10.1016/j.jpain.2006.02.007. PMID 16942948
- [Background] Peuckmann V, Ekholm O, Rasmussen NK, Groenvold M, Christiansen P, Moller S, Eriksen J, Sjogren P. Chronic pain and other sequelae in long-term breast cancer survivors: nationwide survey in Denmark. Eur J Pain. 2009 May;13(5):478-85. doi: 10.1016/j.ejpain.2008.05.015. Epub 2008 Jul 16. PMID 18635381
- [Background] Arman M, Rehnsfeldt A, Lindholm L, Hamrin E. The face of suffering among women with breast cancer-being in a field of forces. Cancer Nurs. 2002 Apr;25(2):96-103. doi: 10.1097/00002820-200204000-00003. PMID 11984096
- [Background] Gartner R, Jensen MB, Nielsen J, Ewertz M, Kroman N, Kehlet H. Prevalence of and factors associated with persistent pain following breast cancer surgery. JAMA. 2009 Nov 11;302(18):1985-92. doi: 10.1001/jama.2009.1568. PMID 19903919
- [Background] Ferlay J, Soerjomataram I, Dikshit R, Eser S, Mathers C, Rebelo M, Parkin DM, Forman D, Bray F. Cancer incidence and mortality worldwide: sources, methods and major patterns in GLOBOCAN 2012. Int J Cancer. 2015 Mar 1;136(5):E359-86. doi: 10.1002/ijc.29210. Epub 2014 Oct 9. PMID 25220842
- [Background] Andersen KG, Kehlet H. Persistent pain after breast cancer treatment: a critical review of risk factors and strategies for prevention. J Pain. 2011 Jul;12(7):725-46. doi: 10.1016/j.jpain.2010.12.005. Epub 2011 Mar 24. PMID 21435953
- [Background] Cheville AL, Tchou J. Barriers to rehabilitation following surgery for primary breast cancer. J Surg Oncol. 2007 Apr 1;95(5):409-18. doi: 10.1002/jso.20782. PMID 17457830
- [Background] Assa J. The intercostobrachial nerve in radical mastectomy. J Surg Oncol. 1974;6(2):123-6. doi: 10.1002/jso.2930060206. No abstract available. PMID 4822897
- [Background] Cunnick GH, Upponi S, Wishart GC. Anatomical variants of the intercostobrachial nerve encountered during axillary dissection. Breast. 2001 Apr;10(2):160-2. doi: 10.1054/brst.2000.0226. PMID 14965578
- [Background] Loukas M, Hullett J, Louis RG Jr, Holdman S, Holdman D. The gross anatomy of the extrathoracic course of the intercostobrachial nerve. Clin Anat. 2006 Mar;19(2):106-11. doi: 10.1002/ca.20226. PMID 16470542
- [Background] Wallace MS, Wallace AM, Lee J, Dobke MK. Pain after breast surgery: a survey of 282 women. Pain. 1996 Aug;66(2-3):195-205. doi: 10.1016/0304-3959(96)03064-3. PMID 8880841
- [Background] Andersen KG, Duriaud HM, Kehlet H, Aasvang EK. The Relationship Between Sensory Loss and Persistent Pain 1 Year After Breast Cancer Surgery. J Pain. 2017 Sep;18(9):1129-1138. doi: 10.1016/j.jpain.2017.05.002. Epub 2017 May 11. PMID 28502878
- [Background] Glare PA, Davies PS, Finlay E, Gulati A, Lemanne D, Moryl N, Oeffinger KC, Paice JA, Stubblefield MD, Syrjala KL. Pain in cancer survivors. J Clin Oncol. 2014 Jun 1;32(16):1739-47. doi: 10.1200/JCO.2013.52.4629. Epub 2014 May 5. PMID 24799477
- [Background] Ahmed A, Bhatnagar S, Rana SP, Ahmad SM, Joshi S, Mishra S. Prevalence of phantom breast pain and sensation among postmastectomy patients suffering from breast cancer: a prospective study. Pain Pract. 2014 Feb;14(2):E17-28. doi: 10.1111/papr.12089. Epub 2013 Jun 24. PMID 23789788
- [Background] Vecht CJ, Van de Brand HJ, Wajer OJ. Post-axillary dissection pain in breast cancer due to a lesion of the intercostobrachial nerve. Pain. 1989 Aug;38(2):171-6. doi: 10.1016/0304-3959(89)90235-2. PMID 2780072
- [Background] Jung BF, Ahrendt GM, Oaklander AL, Dworkin RH. Neuropathic pain following breast cancer surgery: proposed classification and research update. Pain. 2003 Jul;104(1-2):1-13. doi: 10.1016/s0304-3959(03)00241-0. No abstract available. PMID 12855309
- [Background] Macdonald L, Bruce J, Scott NW, Smith WC, Chambers WA. Long-term follow-up of breast cancer survivors with post-mastectomy pain syndrome. Br J Cancer. 2005 Jan 31;92(2):225-30. doi: 10.1038/sj.bjc.6602304. PMID 15655557
- [Background] Leysen L, Beckwee D, Nijs J, Pas R, Bilterys T, Vermeir S, Adriaenssens N. Risk factors of pain in breast cancer survivors: a systematic review and meta-analysis. Support Care Cancer. 2017 Dec;25(12):3607-3643. doi: 10.1007/s00520-017-3824-3. Epub 2017 Aug 10. PMID 28799015
- [Background] Treede RD, Jensen TS, Campbell JN, Cruccu G, Dostrovsky JO, Griffin JW, Hansson P, Hughes R, Nurmikko T, Serra J. Neuropathic pain: redefinition and a grading system for clinical and research purposes. Neurology. 2008 Apr 29;70(18):1630-5. doi: 10.1212/01.wnl.0000282763.29778.59. Epub 2007 Nov 14. PMID 18003941
- [Background] Haroutiunian S, Nikolajsen L, Finnerup NB, Jensen TS. The neuropathic component in persistent postsurgical pain: a systematic literature review. Pain. 2013 Jan;154(1):95-102. doi: 10.1016/j.pain.2012.09.010. PMID 23273105
- [Background] Borsook D, Kussman BD, George E, Becerra LR, Burke DW. Surgically induced neuropathic pain: understanding the perioperative process. Ann Surg. 2013 Mar;257(3):403-12. doi: 10.1097/SLA.0b013e3182701a7b. PMID 23059501
- [Background] Stevens PE, Dibble SL, Miaskowski C. Prevalence, characteristics, and impact of postmastectomy pain syndrome: an investigation of women's experiences. Pain. 1995 Apr;61(1):61-68. doi: 10.1016/0304-3959(94)00162-8. PMID 7644250
- [Background] Jensen MP, Chodroff MJ, Dworkin RH. The impact of neuropathic pain on health-related quality of life: review and implications. Neurology. 2007 Apr 10;68(15):1178-82. doi: 10.1212/01.wnl.0000259085.61898.9e. PMID 17420400
- [Background] Jung BF, Herrmann D, Griggs J, Oaklander AL, Dworkin RH. Neuropathic pain associated with non-surgical treatment of breast cancer. Pain. 2005 Nov;118(1-2):10-4. doi: 10.1016/j.pain.2005.09.014. Epub 2005 Oct 4. No abstract available. PMID 16213086
- [Background] Befort CA, Klemp J. Sequelae of breast cancer and the influence of menopausal status at diagnosis among rural breast cancer survivors. J Womens Health (Larchmt). 2011 Sep;20(9):1307-13. doi: 10.1089/jwh.2010.2308. Epub 2011 Jun 28. PMID 21711155
- [Background] 30. Miale S, Harrington S, Kendig T. Oncology Section Task Force on Breast Cancer Outcomes: Clinical measures of upper extremity function. Rehabil Oncol. 2013;31(1):27-34.
- [Background] Waltho D, Rockwell G. Post-breast surgery pain syndrome: establishing a consensus for the definition of post-mastectomy pain syndrome to provide a standardized clinical and research approach - a review of the literature and discussion. Can J Surg. 2016 Sep;59(5):342-50. doi: 10.1503/cjs.000716. PMID 27668333
- [Background] Chappell AG, Bai J, Yuksel S, Ellis MF. Post-Mastectomy Pain Syndrome: Defining Perioperative Etiologies to Guide New Methods of Prevention for Plastic Surgeons. World J Plast Surg. 2020 Sep;9(3):247-253. doi: 10.29252/wjps.9.3.247. PMID 33329999
- [Background] Perkins FM, Kehlet H. Chronic pain as an outcome of surgery. A review of predictive factors. Anesthesiology. 2000 Oct;93(4):1123-33. doi: 10.1097/00000542-200010000-00038. No abstract available. PMID 11020770
- [Background] Smith WC, Bourne D, Squair J, Phillips DO, Chambers WA. A retrospective cohort study of post mastectomy pain syndrome. Pain. 1999 Oct;83(1):91-5. doi: 10.1016/s0304-3959(99)00076-7. PMID 10506676
- [Background] 35. Keith R. Lohse, PhD, Catherine E. Lang, PT PhD, and Lara A. Boyd PP, Hendrix, Abernethy, Sloane, Misuraca & M. 基因的改变NIH Public Access. Bone. 2013;23(1):1-7.
- [Background] Smith BG, Lewin JS. Lymphedema management in head and neck cancer. Curr Opin Otolaryngol Head Neck Surg. 2010 Jun;18(3):153-8. doi: 10.1097/MOO.0b013e32833aac21. PMID 20463478
- [Background] Schou Bredal I, Smeby NA, Ottesen S, Warncke T, Schlichting E. Chronic pain in breast cancer survivors: comparison of psychosocial, surgical, and medical characteristics between survivors with and without pain. J Pain Symptom Manage. 2014 Nov;48(5):852-62. doi: 10.1016/j.jpainsymman.2013.12.239. Epub 2014 Apr 2. PMID 24703940
- [Background] Andersen KG, Aasvang EK, Kroman N, Kehlet H. Intercostobrachial nerve handling and pain after axillary lymph node dissection for breast cancer. Acta Anaesthesiol Scand. 2014 Nov;58(10):1240-8. doi: 10.1111/aas.12393. PMID 25307709
- [Background] 40. St. Louis MS. Pathology: Implications for the physical therapist. Elsevier..(3rd ed.). 2009.
- [Background] 41. Sleigh BC MB. Lymphedema. InStatPearls [Internet] 2019 . [Internet]. 2019. Available from: https://www.ncbi.nlm.nih.gov/books/NBK537239/
- [Background] 42. Lymphoedema. [Internet]. Physiopedia. 2021. Available from: https://www.physio-pedia.com/Lymphoedema
- [Background] 43. American Cancer Society | Information and Resources about for Cancer: Breast, Colon, Lung, Prostate, Skin. /www.cancer.org/> [Internet]. Cancer.org. 2021. Available from: https://www.cancer.org/
- [Background] 44. April U. Oncology Section EDGE Task Force Report Summaries Colon Cancer Outcomes Authors Urogenital Cancer Outcome Measures. 2018;(August 2015):1-10.
- [Background] Ho K, Spence J, Murphy MF. Review of pain-measurement tools. Ann Emerg Med. 1996 Apr;27(4):427-32. doi: 10.1016/s0196-0644(96)70223-8. No abstract available. PMID 8604852
- [Background] Lowe NK, Walker SN, MacCallum RC. Confirming the theoretical structure of the McGill Pain Questionnaire in acute clinical pain. Pain. 1991 Jul;46(1):53-60. doi: 10.1016/0304-3959(91)90033-T. PMID 1896208
- [Background] De Gagne TA, Mikail SF, D'Eon JL. Confirmatory factor analysis of a 4-factor model of chronic pain evaluation. Pain. 1995 Feb;60(2):195-202. doi: 10.1016/0304-3959(94)00114-T. PMID 7784105
- [Background] Scott J, Huskisson EC. Graphic representation of pain. Pain. 1976 Jun;2(2):175-84. No abstract available. PMID 1026900
- [Background] Gallagher EJ, Liebman M, Bijur PE. Prospective validation of clinically important changes in pain severity measured on a visual analog scale. Ann Emerg Med. 2001 Dec;38(6):633-8. doi: 10.1067/mem.2001.118863. PMID 11719741
- [Background] Jensen MP, Karoly P, Braver S. The measurement of clinical pain intensity: a comparison of six methods. Pain. 1986 Oct;27(1):117-126. doi: 10.1016/0304-3959(86)90228-9. PMID 3785962
- [Background] Jensen MP. The validity and reliability of pain measures in adults with cancer. J Pain. 2003 Feb;4(1):2-21. doi: 10.1054/jpai.2003.1. PMID 14622723
- [Background] Kremer E, Atkinson HJ, Ignelzi RJ. Measurement of pain: patient preference does not confound pain measurement. Pain. 1981 Apr;10(2):241-248. doi: 10.1016/0304-3959(81)90199-8. PMID 7267140
- [Background] Fernandez-Lao C, Cantarero-Villanueva I, Fernandez-de-las-Penas C, Del-Moral-Avila R, Menjon-Beltran S, Arroyo-Morales M. Widespread mechanical pain hypersensitivity as a sign of central sensitization after breast cancer surgery: comparison between mastectomy and lumpectomy. Pain Med. 2011 Jan;12(1):72-8. doi: 10.1111/j.1526-4637.2010.01027.x. Epub 2010 Dec 10. PMID 21143767
- [Background] Jensen MP, Turner JA, Romano JM. What is the maximum number of levels needed in pain intensity measurement? Pain. 1994 Sep;58(3):387-392. doi: 10.1016/0304-3959(94)90133-3. PMID 7838588
- [Background] Jensen MP, Turner JA, Romano JM, Fisher LD. Comparative reliability and validity of chronic pain intensity measures. Pain. 1999 Nov;83(2):157-62. doi: 10.1016/s0304-3959(99)00101-3. PMID 10534586